CLINICAL TRIAL: NCT00117182
Title: A Phase II Study to Investigate Mannitol Challenge as a Tool to Predict Treatment Response to Inhaled Corticosteroids in COPD
Brief Title: Aridol Challenge as a Tool to Predict Treatment Response to Inhaled Corticosteroids in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DPM-COPD-201
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Lung Diseases, Obstructive
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Budesonide; Ipratropium; Albuterol

INTERVENTIONS:
Drug: Dry powder mannitol
Drug: Budesonide 400mcg administered via turbuhaler
Drug: Ipratropium bromide 80mcg
Drug: Salbutamol 400mcg

SUMMARY:
The purpose of this study is to determine whether the Aridol (mannitol) challenge test can predict response to treatment with inhaled corticosteroids in COPD subjects. Subjects will undergo an Aridol test and then 3 months of treatment with inhaled corticosteroids. The effect on lung function and quality of life will then be measured and correlated with the Aridol test result.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (history, spirometry, symptoms including chronic cough and/or shortness of breath that is worse on exertion and/or excess sputum production)
* Aged 45 - 80 years
* Have pre-bronchodilator FEV1 > 1.4 litres and at least 60% of predicted for height, age and gender and a post-bronchodilator FEV1 <80% of predicted for height, age and gender
* Post-bronchodilator FEV1/FVC < 70 %
* ≥ 10 pack years smoking history
* As determined by the investigator, are capable and willing to:

  * perform all of the techniques necessary to measure lung function;
  * administer the dry powder mannitol.
* Are capable of, and have given informed consent to, participating in this study in accordance with local regulations.
* The subject must be in stable clinical condition at the time of, and for a period of 14 days prior to, their recruitment into the study. Stable clinical condition is defined as lack of:

  * change in sputum production (volume, colour, consistency);
  * increased cough;
  * worsening dyspnoea;
  * increased malaise, fatigue or lethargy;
  * reduction in exercise tolerance;
  * fever;
  * antibiotic treatment (for respiratory infection).

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted.
* Subjects receiving treatment with inhaled corticosteroids (including combination therapies, e.g. Seretide®, Symbicort®) or oral corticosteroids within the last 6 weeks.
* Subjects who have had an exacerbation or a chest infection within the 2 weeks prior to the study.
* Subjects receiving antibiotic treatment for respiratory infection.
* Known diagnosis of asthma or allergic rhinitis.
* Myocardial infarction in the six months prior to enrolment.
* Cerebral vascular accident in the six months prior to enrolment.
* Ocular surgery in the three months prior to enrolment.
* Abdominal surgery in the three months prior to enrolment.
* Active tuberculosis (TB).
* Lung cancer or any other malignancies, which are considered by the investigator as a contraindication to participating in the study.
* Lung disease other than COPD (e.g. bronchiectasis).
* Uncontrolled insulin-dependant or non-insulin dependant diabetes, i.e. >10% HbA1c.
* Female subjects of reproductive capability, not using a reliable form of contraception
* Inability to obtain informed consent from the subject or subject's authorised representative.
* Subjects who have participated in another investigative drug study parallel to, or within 4 weeks of, study entry.
* Known intolerance to mannitol.
* Uncontrolled hypertension - systolic blood pressure (BP) > 200 mmHg and or diastolic BP > 100 mmHg.
* Planned pulmonary rehabilitation.
* Have had major abdominal, chest or brain surgery in the three months prior to enrolment.
* Have known cerebral, aortic or abdominal aneurysm.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2005-07; Study Completion 2006-08

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1)

SECONDARY OUTCOMES:
Response dose ratio (RDR)
Dose of provoking stimulus causing a 15%, 12% or 10% fall in FEV1 (PD15, PD12, PD10)
Lung function values
Quality of life assessed by St. George's Respiratory Questionnaire (SGRQ)- total score
COPD clinical control scores (CCQ)
Exacerbation frequency
Days on antibiotics
Days off work or days unable to carry out normal activities
Reversibility of airflow obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Ing, MBBS, Principal Investigator — Bankstown Hospital; Martin Coffey, MBBS, Principal Investigator — Rosebud Medical Centre; David Langton, MBBS, Principal Investigator — Peninsula Chest Clinic, Frankston; Chris Steinfort, MBBS, Principal Investigator — The Rooms of Dr Steinfort, Geelong; Trevor WIlliams, MBBS, Principal Investigator — The Alfred; Peter Frith, MBBS, Principal Investigator — Flinders Medical Centre; Michael Chia, MBBS, Principal Investigator — Respiratory Research Foundation, Toorak Gardens; Maureen McKeirnan, MBBS, Principal Investigator — Brisbane South Medical Centre; Fred de Looze, MBBS, Principal Investigator — Centre for General Practice for Clinical Trials Unit, Inala; Michael Crookes, MBBS, Principal Investigator — Peninsula Medical Centre; Alan James, MBBS, Principal Investigator — Sir Charles Gairdner Hospital; Phillip Thompson, MBBS, Principal Investigator — Mount Medical Centre
Locations (13):
- Australia (13):
  - Respiratory Clinic, Sydney, New South Wales
  - Peninsula Medical Centre, Umina, New South Wales
  - Wesley Medical Centre, Auchenflower, Queensland
  - Brisbane South Clinical Clinical Research Centre, Brisbane, Queensland
  - Inala Health Centre, PO BOx 52, Inala, Queensland
  - Flinders University, Bedford Park, South Australia
  - Respiratory Research Foundation Clinical Trial Centre, Toorak Gardens, South Australia
  - Peninsula Chest Clinic, Frankston, Victoria
  - The rooms of Dr Chris Steinfort, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Rosebud Medical Centre, Rosebud, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Mount Medical Centre, Perth, Western Australia

REFERENCES:
- [Background] Anderson SD, Brannan J, Spring J, Spalding N, Rodwell LT, Chan K, Gonda I, Walsh A, Clark AR. A new method for bronchial-provocation testing in asthmatic subjects using a dry powder of mannitol. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):758-65. doi: 10.1164/ajrccm.156.3.9701113. PMID 9309990
- [Background] Brannan JD, Koskela H, Anderson SD, Chan HK. Budesonide reduces sensitivity and reactivity to inhaled mannitol in asthmatic subjects. Respirology. 2002 Mar;7(1):37-44. doi: 10.1046/j.1440-1843.2002.00357.x. PMID 11896899
- [Background] Burge PS, Calverley PM, Jones PW, Spencer S, Anderson JA. Prednisolone response in patients with chronic obstructive pulmonary disease: results from the ISOLDE study. Thorax. 2003 Aug;58(8):654-8. doi: 10.1136/thorax.58.8.654. PMID 12885977
- [Background] Koskela HO, Hyvarinen L, Brannan JD, Chan HK, Anderson SD. Sensitivity and validity of three bronchial provocation tests to demonstrate the effect of inhaled corticosteroids in asthma. Chest. 2003 Oct;124(4):1341-9. doi: 10.1378/chest.124.4.1341. PMID 14555564
- [Background] Leuppi JD, Tandjung R, Anderson SD, Stolz D, Brutsche MH, Bingisser R, Perruchoud AP, Surber C, Knoblauch A, Andersson M, Greiff L, Chan HK, Tamm M. Prediction of treatment-response to inhaled corticosteroids by mannitol-challenge test in COPD. A proof of concept. Pulm Pharmacol Ther. 2005;18(2):83-8. doi: 10.1016/j.pupt.2004.10.005. Epub 2004 Dec 21. PMID 15649849